CLINICAL TRIAL: NCT06797297
Title: A Phase II, Open-label, Randomized, Multi-center Study to Evaluate the Efficacy and Safety of IBI363 Monotherapy Compared to Pembrolizumab in Patients With Unresectable Locally Advanced or Metastatic Mucosal and Acral Melanoma Who Had Not Previously Received Systemic Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of IBI363 Monotherapy Compared to Pembrolizumab in Patients With Unresectable Locally Advanced or Metastatic Mucosal or Acral Melanoma Who Had Not Previously Received Systemic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363B202
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Participants are assigned to one of two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: IBI363 (Experimental)
  Interventions: Biological: IBI363
- Active Comparator: Pembrolizumab (Active Comparator)
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: IBI363 — a mutated IL-2 cytokine fused to an anti-PD-1 antibody to combine IL-2 pathway stimulation with checkpoint blockade.
  Arms: Experimental: IBI363
Biological: Pembrolizumab — Pembrolizumab is a humanized monoclonal anti-PD1 antibody
  Arms: Active Comparator: Pembrolizumab

SUMMARY:
This is a Phase II, open-label, randomized, multi-center study to assess the efficacy and safety of IBI363 monotherapy compared to Pembrolizumab in the treatment of patients with unresectable locally advanced or metastatic mucosal or acral melanoma who had not previously received systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable, locally advanced or metastatic mucosal or acral-type melanoma, according to the American Joint Committee on Cancer (AJCC) 8th edition stage III-IV.
2. No prior systemic treatment for unresectable or metastatic melanoma; Prior adjuvant or neoadjuvant therapy (except for disease progression to unresectable or metastatic melanoma during adjuvant or neoadjuvant therapy or within 6 months after treatment discontinuation) was permitted.
3. Have at least one measurable lesion (target lesion) according to RECIST v1.1. For lesions that have previously received radiotherapy or intratumoral injection, measurable lesions that progress to the criteria specified in RECIST1.1 after treatment may be considered.

   The target lesions of this study must be measured by imaging (enhanced CT or MRI. Plain scan CT or MRI can be accepted after communication with the sponsor if the subjects are allergic to contrast media or have other conditions that are not suitable for enhanced CT or MRI).

   Skin lesions or other superficial sites that cannot be repeatedly measured by imaging can only be used as non-target lesions.
4. The Eastern Cooperative Oncology Group Physical Status Score (ECOG PS) is 0 or 1.
5. Expected survival time no less than 3 months.
6. Female subjects of childbearing age or male subjects whose partner is a female of childbearing age agree to strictly use effective contraception throughout the treatment period and for 6 months after the treatment period.
7. Breastfeeding women must agree to strictly refrain from breastfeeding during the entire treatment period and for 6 months after the treatment period.

Exclusion Criteria:

1. Women who are pregnant or plan to become pregnant within 6 months before, during, or after the last dose of the study drug.
2. Active or symptomatic central nervous system metastases
3. Any of the following hematological abnormalities were present at baseline * (within 7 days before the first administration of the study drug) :

   Hemoglobin <90 g/L The absolute count of neutrophils (ANC) was <1.5×10^9/L Platelet count <100×10^9/L
4. Any of the following serum biochemical abnormalities are present at baseline (within 7 days before the first dose) :

   Total bilirubin >1.5× Upper limit of normal (ULN); Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3×ULN; For liver metastasis, AST or ALT > 5.0×ULN; With serum Creatinine >1.5×ULN or Clearance of Creatinine (CCr) <45 mL/min, CCr (using actual body weight) was calculated using Cockcroft-Gault formula (Appendix 3).

   Albumin <30 g/L.
5. Any of the following coagulation parameters are abnormal at baseline (within 7 days before the first dose) :

   International normalizaed ratio (INR) >1.5×ULN (>3×ULN if receiving steady dose anticoagulant therapy); Partial thromboplastin time (PTT) (or activated partial thromboplastin time, [activated partial thromboplastin time, PTT) aPTT]) >1.5×ULN (>3×ULN if receiving steady dose anticoagulant therapy).
6. There is a history of active thrombosis or deep vein thrombosis or pulmonary embolism in the 4 weeks prior to initial administration of the investigatory drug, unless the disease is adequately treated and is considered stable by the investigator.
7. Uncontrolled bleeding or a known tendency to bleed.
8. Cardiovascular and cerebrovascular diseases of significant clinical significance.
9. History of interstitial pneumonia, pulmonary fibrosis, pneumoconiosis, drug-related pneumonia, radiation pneumonia, etc. requiring steroid hormone or other treatment, as well as severe abnormal lung function or other forms of restrictive lung disease.
10. An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, corticosteroids, or immunosuppressants) has occurred within 2 years prior to first administration. Replacement therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
IRRC-Progression Free Survival(PFS) | up to 2 years
  Progression Free Survival assessed by Independent Radiology Review Committee (IRRC-PFS), Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
INV-Progression Free Survival(PFS) | up to 2 years
  Progression Free Survival assessed by Investigator, Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Objective Response Rate (ORR) | up to 2 years
  Objective response rate (ORR) in two arms based on RECIST V1.1 by IRRC and investigator.
Duration of Response (Duration Of Response) | up to 2 years
  DOR in two arms based on RECIST V1.1 by IRRC and investigator.
Disease Control Rate (DCR) | up to 2 years
  DCR in two arms based on RECIST V1.1 by IRRC and investigator.
Time to Response (TTR) | up to 2 years
  TTR in two arms based on RECIST V1.1 by IRRC and investigator.
Overall Survival (OS) | up to 2 years
  Overall survival in two arms
safety indicators during the treatment | up to 2 years
  Number of participants with Adverse Event (AE), Treatment Emergent Adverse Event (TEAE), Immune-related AE (irAE), Serious Adverse Event (SAE), treatment-emergent AE leading to treatment termination, death, and related with investigational agent

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Jishuitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, China,, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Third people's hospital of Zhengzhou, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Hena
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Second Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Baotou Cancer Hospital, Baotou, Inner Mongolia
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No